CLINICAL TRIAL: NCT04190134
Title: Development of a Behavioral Intervention With Socially Assistive Robots to Enhance Magnification Device Use for Reading
Brief Title: Socially Assistive Robots to Enhance Magnification Device Use for Reading
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Ava K. Bittner, OD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-001429
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Low Vision
Keywords: robot
MeSH Terms: conditions — Vision, Low | interventions — Robotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Robot (Experimental): One month after study entry, participants will receive the robot at home for two months, followed by a three month observation period without the robot.
  Interventions: Behavioral: Socially Assistive Robot for Low Vision Rehabilitation
- Delayed/Waitlist Robot (Active Comparator): Three months after study entry, participants will receive the robot at home for three months.
  Interventions: Behavioral: Socially Assistive Robot for Low Vision Rehabilitation

INTERVENTIONS:
Behavioral: Socially Assistive Robot for Low Vision Rehabilitation — A socially assistive robot will be customized to engage in dialog and conversations to motivate and encourage optimal use of new magnification devices for reading at home by individuals with vision loss.

SUMMARY:
The aims of this exploratory research project are to customize, deploy and evaluate the preliminary efficacy of a socially assistive robot as a novel approach to motivate and encourage optimal, long-term use of new magnification devices for reading in individuals with vision loss. The goals are to promote patient acceptance, adherence and skills reinforcement to achieve proficiency in the use of the magnifier, in order to attempt to reduce visual disability while performing important daily activities, such as reading tasks. This is a high priority given the increasing prevalence of low vision, paucity of low vision rehabilitation providers, and barriers related to access to care, such as transportation and geography, all of which motivate the development of this complementary approach for the provision of additional support at home by the socially assistive robot.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with any level of vision loss due to any ocular disease,
* age 18 and older,
* received a magnification device(s) (i.e., hand-held optical magnifiers, portable electronic video magnifiers, some stand magnifiers and CCTVs) from the UCLA Vision Rehabilitation Center.

Exclusion Criteria:

* schedules not permitting participation in planned study sessions or visits (including planning to move or take extended vacation during study period),
* inability to understand study procedures or communicate responses to visual stimuli in a consistent manner (cognitive impairment as per TICS),
* substance abuse,
* significant hearing loss (unable to hear communication by phone or from robot),
* significant medical condition likely to limit participation or lifespan,
* their magnifier device has features that would not work in conjunction with the beacon sensors: (1) hands-free and do not have a place where the patient's hand is holding the device during use (therefore, they would not register a significant change in temperature), and/or (2) no surface area of at least 1"x1" to which the beacon sensor could be attached without interfering with the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Activity Inventory | change from 1 month post-enrollment to 2-3 months after receiving the socially assistive robot
  questionnaire; scores will be Rasch analyzed in logic units with higher or positive scores indicating less difficulty (i.e., improvement)

SECONDARY OUTCOMES:
MNread | For Immediate robot: baseline, 1 month, 3 months, 6 months. For Delayed/Waitlist robot: baseline, 3 months, 6 months.
  reading test
Sustained Silent Reading Test | baseline and monthly for 6 months
  reading test
Geriatric Depression Scale (GDS) | baseline and monthly for 6 months
  questionnaire; scale ranges from 0 to 15 with higher values indicating greater depression
PANAS | baseline and monthly for 6 months
  questionnaire; scale ranges from 10 to 50 with higher values indicating greater positive moods
Perceived Stress Scale | baseline and monthly for 6 months
  questionnaire; scale ranges from 0 to 56 with higher values indicating greater perceived stress
3-item UCLA Loneliness Scale | baseline and monthly for 6 months
  questionnaire; scale ranges from 3 to 9 with higher values indicating greater loneliness
Duke Social Support Index | baseline and monthly for 6 months
  questionnaire; scale ranges from 10 to 30 with higher values indicating greater social support
Almere | 1 month post-enrollment and 2-3 months after receiving the socially assistive robot
  questionnaire; scale ranges from 41 to 205 with higher values indicating greater acceptance of robots

CONTACTS AND LOCATIONS:
Overall Officials: Ava K Bittner, OD, PhD, Principal Investigator — UCLA Stein Eye Institute; Vision Rehabilitation Center; Maja J Mataric, PhD, Principal Investigator — USC Interaction Lab; Viterbi School of Engineering
Locations (1):
- UCLA Stein Eye Institute, Los Angeles, California, United States